CLINICAL TRIAL: NCT03122821
Title: Effect of Transcranial Stimulation Augmented With Mental Imagery in Upper Limb Stroke Rehabilitation: A Randomized Controlled Trial
Brief Title: Trans Cranial Brain Stimulation for Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Majmaah University (Other)
Responsible Party: Principal Investigator, faizan kashoo, PT, Principal Investigator, Majmaah University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MajmaahU
Record Dates: First submitted 2017-04-13; First posted 2017-04-21 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Transcranial magnetic stimulation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: transcranial electrical stimulation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Real Trans-cranial direct stimulation + Mental Imagery
  Interventions: Other: Real Transcranial direct stimulation+Mental Imagery
- Group 2 (Active Comparator): Sham Trans-cranial direct stimulation + Mental imagery
  Interventions: Other: Sham Transcranial Direct Stimulation +Mental Imagery

INTERVENTIONS:
Other: Real Transcranial direct stimulation+Mental Imagery — The subject will be practicing mental imagery along with mental imagery. A video of the task will be played in front of the patient and the subject will be asked to perform the mental practice of the activity.The video will be played thrice.The electrodes will be placed at the premotor cortex over the scalp corresponding to the topographical representation of upper limb on the contralateral cerebral hemisphere.Transcranial direct current stimulation (tDCS), (or "Transcranial Micropolarization"), is the most commonly used type of tCS [2, 19-25]. It employs a battery-driven stimulator to deliver weak direct currents (1.5 mA) through contact electrodes over the scalp. The current flow modulates neuronal excitability by altering the resting membrane potential of the neurons and produces aftereffects.Transcranial magnetic stimulation for 30 minutes, 5 days a week for 2 weeks.Transcranial direct stimulation for 30 minutes, 5 days a week for 2 weeks
  Arms: Group 1
Other: Sham Transcranial Direct Stimulation +Mental Imagery — The electrodes will be placed at the premotor cortex over the scalp corresponding to the topographical representation of upper limb on the contralateral cerebral hemisphere.Transcranial direct current stimulation (tDCS), (or "Transcranial Micropolarization"), is the most commonly used type of tCS [2, 19-25]. It employs a battery-driven stimulator to deliver weak direct currents (1.5 mA) through contact electrodes over the scalp. The current flow modulates neuronal excitability by altering the resting membrane potential of the neurons and produces aftereffects.Transcranial magnetic stimulation for 30 minutes, 5 days a week for 2 weeks.Transcranial direct stimulation for 30 minutes, 5 days a week for 2 weeks
  Arms: Group 2

SUMMARY:
Noninvasive brain stimulation (NIBS) refers to a group of modalities that are used to induce electric currents to and within the brain for diagnostic or therapeutic purposes. Two major types of NIBS techniques are currently in use on humans for clinical and research applications: Transcranial Magnetic Stimulation (TMS) and Transcranial Current Stimulation (tCS). Moreover, the studies evaluating the clinical benefit of mental practice in stroke so far are mostly small feasibility studies, while the few randomized controlled trials reported had relatively small sample sizes. As such, the evidence for mental practice in the treatment of movement disorders following stroke, and other neurological conditions, remains somewhat anecdotal. Purpose of our research is to show the effect of combining brain stimulation and mental imagery on functional recovery of upper limb in stroke.

DETAILED DESCRIPTION:
TITLE Effect of Transcranial Stimulation augmented with Mental Imagery in Upper Limb Stroke Rehabilitation: A Randomized Controlled Trial

Mr. Faizan Zaffar Kashoo

Department of Physical Therapy and Health rehabilitation, College of Applied Medical sciences. Majmaah University. KSA

INTRODUCTION

Noninvasive brain stimulation (NIBS) refers to a group of modalities that are used to induce electric currents to and within the brain for diagnostic or therapeutic purposes [1-4]. A growing body of evidence suggests that NIBS techniques may have a promising role in the diagnosis, monitoring, and treatment of a variety of neurological and psychiatric conditions [5-9]. The therapeutic potential of NIBS stems from the capacity to evoke immediate and sustained modulation of neural network activity through alterations in neuronal excitation. The induced neuromodulation can be either excitatory or inhibitory, depending on the polarity, frequency, and duration of the stimulation [2, 10]. Moreover, the ability to induce directional modulation further enhances the therapeutic possibilities of NIBS, as the necessary direction of the brain excitability for recovery varies with different disease conditions [10, 11].

Two major types of NIBS techniques are currently in use on humans for clinical and research applications: Transcranial Magnetic Stimulation (TMS) and Transcranial Current Stimulation (tCS) [12]. TMS uses a varying magnetic field to induce weak electric currents in the brain. It can be delivered as a single pulse or as a train of pulses. Single-pulse TMS is typically used to study brain physiology and plasticity [3, 13-16], whereas repetitive-pulse TMS (rTMS) is commonly used to elicit neuromodulation and neuroplasticity, and can result in prolonged excitability changes that outlast the stimulation period [6, 15]. Typically, the direction of neuromodulation is driven by the frequency at which the stimulation is performed, such that high-frequency rTMS increases cortical excitability and low-frequency rTMS decreases cortical excitability [17]. However, theta burst stimulation (a variation of high frequency rTMS) can induce either depression or facilitation of cortical excitability, depending on burst-train duration, such that intermittent theta burst stimulation increases cortical excitability and continuous theta burst stimulation decreases cortical excitability [18].

tCS refers to the application of direct or alternating current on a specific region of the brain, transmitted via electrodes attached to the scalp. A wide range of tCS modalities exists, but only a few have been well-studied. Transcranial direct current stimulation (tDCS), (or "Transcranial Micropolarization"), is the most commonly used type of tCS [2, 19-25]. It employs a battery-driven stimulator to deliver weak direct currents (0.5-2.0 mA) through contact electrodes over the scalp. The current flow modulates neuronal excitability by altering the resting membrane potential of the neurons and produces aftereffects (i.e., prolonged changes in neuronal excitability) that are thought to be driven by Glutamatergic and GABAergic synapsic plasticity [26]. tDCS can be used to elicit an excitatory (anodal) or inhibitory (cathodal) effect, depending on the polarity of stimulation. Specifically, anodal stimulation has a depolarizing effect, which increases neuronal excitability; whereas, cathodal stimulation has a hyperpolarizing effect, which decreases neuronal excitability [1, 19, 27, 28].

Much interest has been raised by the potential of mental practice of motor tasks, also called 'motor imagery', as a neuro-rehabilitation technique to enhance motor recovery following stroke 29-31. The appeal of motor imagery as a potentially effective neuro-rehabilitation technique is popular, which is reflected in multiple reviews of relatively few reported clinical evaluations. Moreover, the studies evaluating the clinical benefit of mental practice in stroke so far are mostly small feasibility studies, while the few randomized controlled trials reported had relatively small sample sizes. As such, the evidence for mental practice in the treatment of movement disorders following stroke, and other neurological conditions, remains somewhat anecdotal. Purpose of our research is to show the effect of combined effect of brain stimulation and mental imagery.

RESEARCH HYPOTHESIS

There will be a significant difference between control and experimental groups.

NULL HYPOTHESIS

There will be no significant difference between control and experimental groups.

STUDY DESIGN (TYPE OF STUDY)

Doubled blinded randomized controlled trial.

STUDY POPULATION AND SAMPLING

Chronic stroke and random sampling

DATA COLLECTION METHODS AND INSTRUMENTS

Procedure:

The electrodes will be placed at the premotor cortex over the scalp corresponding to the topographical representation of upper limb on the contralateral cerebral hemisphere.

Transcranial direct stimulation for 30 minutes, 5 days a week for 2 weeks Mental imagery as visual imagery shown to the patient with the help of videotape.

Instrumentation:

Fugl Meyers Scale ARAT

Activities:

exercises: 1. stacking blocks; 2. flipping scrapbook pages; 3. nine-hole pegboard; 4. grabbing saucepan and pouring water into a cup; and 5. opening hand to grasp and pick up cup.

DATA ANALYSIS METHODS

An appropriate quantitative statistical method will be used

STUDY PERIOD

2 year

ELIGIBILITY:
Inclusion Criteria:

1. Having stroke past 6 months.

Exclusion Criteria:

1. Subarachnoid hemorrhage
2. Prior to stroke resulting in aphasia
3. Brain surgery in the past
4. Epileptic activity in the past 12 months
5. Premorbid (suspected) dementia
6. Premorbid psychiatric disease affecting communication (for example, personality disorder)
7. Excessive use of alcohol or drugs
8. Presence of a cardiac pacemaker
9. Metal implants

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Fugl Meyers scale for upper limb | 15 minutes
  Subjects will be rated on impairment of upper limb. The maximum score of 66 for the upper limb, higher scores imply better outcomes.

SECONDARY OUTCOMES:
Action research Arm Test | 15 minutes
  Subjects will be rated on performance and functional activity. The maximum score of 56 for the upper limb, higher scores imply better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Faizan Z Kashoo, Masters, Principal Investigator — Majmaah University
Locations (1):
- NIIMS University hospital, Jaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guleyupoglu B, Schestatsky P, Edwards D, Fregni F, Bikson M. Classification of methods in transcranial electrical stimulation (tES) and evolving strategy from historical approaches to contemporary innovations. J Neurosci Methods. 2013 Oct 15;219(2):297-311. doi: 10.1016/j.jneumeth.2013.07.016. Epub 2013 Aug 14. PMID 23954780
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Kobayashi M, Pascual-Leone A. Transcranial magnetic stimulation in neurology. Lancet Neurol. 2003 Mar;2(3):145-56. doi: 10.1016/s1474-4422(03)00321-1. PMID 12849236
- [Background] Eldaief MC, Press DZ, Pascual-Leone A. Transcranial magnetic stimulation in neurology: A review of established and prospective applications. Neurol Clin Pract. 2013 Dec;3(6):519-526. doi: 10.1212/01.CPJ.0000436213.11132.8e. PMID 24353923
- [Background] Paulus W, Peterchev AV, Ridding M. Transcranial electric and magnetic stimulation: technique and paradigms. Handb Clin Neurol. 2013;116:329-42. doi: 10.1016/B978-0-444-53497-2.00027-9. PMID 24112906
- [Background] Webster BR, Celnik PA, Cohen LG. Noninvasive brain stimulation in stroke rehabilitation. NeuroRx. 2006 Oct;3(4):474-81. doi: 10.1016/j.nurx.2006.07.008. PMID 17012061
- [Background] Radhu N, de Jesus DR, Ravindran LN, Zanjani A, Fitzgerald PB, Daskalakis ZJ. A meta-analysis of cortical inhibition and excitability using transcranial magnetic stimulation in psychiatric disorders. Clin Neurophysiol. 2013 Jul;124(7):1309-20. doi: 10.1016/j.clinph.2013.01.014. Epub 2013 Feb 26. PMID 23485366
- [Background] Edwards MJ, Talelli P, Rothwell JC. Clinical applications of transcranial magnetic stimulation in patients with movement disorders. Lancet Neurol. 2008 Sep;7(9):827-40. doi: 10.1016/S1474-4422(08)70190-X. PMID 18703005
- [Background] Nitsche MA, Paulus W. Noninvasive brain stimulation protocols in the treatment of epilepsy: current state and perspectives. Neurotherapeutics. 2009 Apr;6(2):244-50. doi: 10.1016/j.nurt.2009.01.003. PMID 19332316
- [Background] Boggio PS, Nunes A, Rigonatti SP, Nitsche MA, Pascual-Leone A, Fregni F. Repeated sessions of noninvasive brain DC stimulation is associated with motor function improvement in stroke patients. Restor Neurol Neurosci. 2007;25(2):123-9. PMID 17726271
- [Background] Davis NJ, van Koningsbruggen MG. "Non-invasive" brain stimulation is not non-invasive. Front Syst Neurosci. 2013 Dec 23;7:76. doi: 10.3389/fnsys.2013.00076. eCollection 2013. No abstract available. PMID 24391554
- [Background] Krishnan C, Dhaher Y. Corticospinal responses of quadriceps are abnormally coupled with hip adductors in chronic stroke survivors. Exp Neurol. 2012 Jan;233(1):400-7. doi: 10.1016/j.expneurol.2011.11.007. Epub 2011 Nov 15. PMID 22116042
- [Background] Krishnan C, Ranganathan R, Kantak SS, Dhaher YY, Rymer WZ. Active robotic training improves locomotor function in a stroke survivor. J Neuroeng Rehabil. 2012 Aug 20;9:57. doi: 10.1186/1743-0003-9-57. PMID 22906099
- [Background] Pascual-Leone A, Tormos JM, Keenan J, Tarazona F, Canete C, Catala MD. Study and modulation of human cortical excitability with transcranial magnetic stimulation. J Clin Neurophysiol. 1998 Jul;15(4):333-43. doi: 10.1097/00004691-199807000-00005. PMID 9736467
- [Background] Madhavan S, Krishnan C, Jayaraman A, Rymer WZ, Stinear JW. Corticospinal tract integrity correlates with knee extensor weakness in chronic stroke survivors. Clin Neurophysiol. 2011 Aug;122(8):1588-94. doi: 10.1016/j.clinph.2011.01.011. Epub 2011 Feb 17. PMID 21333591
- [Background] Peterchev AV, Wagner TA, Miranda PC, Nitsche MA, Paulus W, Lisanby SH, Pascual-Leone A, Bikson M. Fundamentals of transcranial electric and magnetic stimulation dose: definition, selection, and reporting practices. Brain Stimul. 2012 Oct;5(4):435-53. doi: 10.1016/j.brs.2011.10.001. Epub 2011 Nov 1. PMID 22305345
- [Background] Mix A, Benali A, Eysel UT, Funke K. Continuous and intermittent transcranial magnetic theta burst stimulation modify tactile learning performance and cortical protein expression in the rat differently. Eur J Neurosci. 2010 Nov;32(9):1575-86. doi: 10.1111/j.1460-9568.2010.07425.x. Epub 2010 Oct 18. PMID 20950358
- [Background] Nitsche MA, Cohen LG, Wassermann EM, Priori A, Lang N, Antal A, Paulus W, Hummel F, Boggio PS, Fregni F, Pascual-Leone A. Transcranial direct current stimulation: State of the art 2008. Brain Stimul. 2008 Jul;1(3):206-23. doi: 10.1016/j.brs.2008.06.004. Epub 2008 Jul 1. PMID 20633386
- [Background] Nitsche MA, Liebetanz D, Lang N, Antal A, Tergau F, Paulus W. Safety criteria for transcranial direct current stimulation (tDCS) in humans. Clin Neurophysiol. 2003 Nov;114(11):2220-2; author reply 2222-3. doi: 10.1016/s1388-2457(03)00235-9. No abstract available. PMID 14580622
- [Background] Nitsche MA, Nitsche MS, Klein CC, Tergau F, Rothwell JC, Paulus W. Level of action of cathodal DC polarisation induced inhibition of the human motor cortex. Clin Neurophysiol. 2003 Apr;114(4):600-4. doi: 10.1016/s1388-2457(02)00412-1. PMID 12686268
- [Background] Nitsche MA, Paulus W. Sustained excitability elevations induced by transcranial DC motor cortex stimulation in humans. Neurology. 2001 Nov 27;57(10):1899-901. doi: 10.1212/wnl.57.10.1899. PMID 11723286
- [Background] Bogdanov OV, Pinchuk DYu, Pisar'kova EV, Shelyakin AM, Sirbiladze KT. The use of the method of transcranial micropolarization to decrease the severity hyperkineses in patients with infantile cerebral palsy. Neurosci Behav Physiol. 1994 Sep-Oct;24(5):442-5. doi: 10.1007/BF02359800. No abstract available. PMID 7838369
- [Background] Ilyukhina VA, Kozhushko NY, Matveev YK, Ponomareva EA, Chernysheva EM, Shaptilei MA. Transcranial micropolarization in the combined therapy of speech and general psychomotor retardation in children of late preschool age. Neurosci Behav Physiol. 2005 Nov;35(9):969-76. doi: 10.1007/s11055-005-0153-7. PMID 16270180
- [Background] Shelyakin AM, Preobrazhenskaya IG, Kassil' MV, Bogdanov OV. The effects of transcranial micropolarization on the severity of convulsive fits in children. Neurosci Behav Physiol. 2001 Sep-Oct;31(5):555-60. doi: 10.1023/a:1010487201282. PMID 11693481
- [Background] Stagg CJ, Nitsche MA. Physiological basis of transcranial direct current stimulation. Neuroscientist. 2011 Feb;17(1):37-53. doi: 10.1177/1073858410386614. PMID 21343407
- [Background] Arul-Anandam AP, Loo C, Sachdev P. Transcranial direct current stimulation - what is the evidence for its efficacy and safety? F1000 Med Rep. 2009 Jul 27;1:58. doi: 10.3410/M1-58. PMID 20948722
- [Background] Krishnan C, Ranganathan R, Kantak SS, Dhaher YY, Rymer WZ. Anodal transcranial direct current stimulation alters elbow flexor muscle recruitment strategies. Brain Stimul. 2014 May-Jun;7(3):443-50. doi: 10.1016/j.brs.2014.01.057. Epub 2014 Jan 29. PMID 24582369
- [Background] Altschuler EL, Wisdom SB, Stone L, Foster C, Galasko D, Llewellyn DM, Ramachandran VS. Rehabilitation of hemiparesis after stroke with a mirror. Lancet. 1999 Jun 12;353(9169):2035-6. doi: 10.1016/s0140-6736(99)00920-4. No abstract available. PMID 10376620
- [Background] Annett J. Motor imagery: perception or action? Neuropsychologia. 1995 Nov;33(11):1395-417. doi: 10.1016/0028-3932(95)00072-b. PMID 8584177
- [Background] Barsalou LW. Grounded cognition. Annu Rev Psychol. 2008;59:617-45. doi: 10.1146/annurev.psych.59.103006.093639. PMID 17705682